CLINICAL TRIAL: NCT04944329
Title: Association Between Covid-19 Disease and Mortality After Hip Fracture Surgery in Elderly: a Multicentre National French Survey
Brief Title: Hip Fracture and COVID-19
Acronym: COLCOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/PC-02
Record Dates: First submitted 2021-06-26; First posted 2021-06-29 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV2 Infection; Hip Fractures; Surgery
MeSH Terms: conditions — COVID-19; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COLCOVID: adults undergoing hip fracture surgery
  Interventions: Procedure: Hip fracture surgery

INTERVENTIONS:
Procedure: Hip fracture surgery — Hip fracture surgery

SUMMARY:
Hip fracture in the elderly is a worldwide public health issue and a medical challenge for early postoperative rehabilitation. More than 2 million people are treated annually with an annual incidence between 100 and 300/100,000 (USA, Europe, China), resulting in a cost of billion dollars and a strain on most surgical facilities. In this context, an early surgical management of patient with fracture within the first 24-48h has been shown to reduce morbidity, length of hospital stay and mortality.

During the Covid-19 pandemics, a higher risk of 30-day mortality has been reported in patients with pre-operative SARS-CoV-2 infection diagnosed 0-2 weeks, 3-4 weeks and 5-6 weeks before surgery compared with patients who did not have a pre-operative SARS-CoV-2 infection. However, this risk seems to disappear in patients diagnosed with SARS-CoV-2 ≥ 7 weeks before surgery. These findings led to propose delayed elective surgery when the benefit-risk ratio was acceptable (cancer, cardiac surgeries). However, delaying surgery in COVID-19 patients (with high risk of immune and thrombotic disorders) with hip fracture could be questionable as the risk related to COVID-19 could be counteracted by the risk delayed surgery.

For assessing the mortality risk related to hip fracture surgery associated with COVID-19, we decided to use the French national hospital discharge records database for comparing the 30-day postoperative mortality in patients with hip fracture and with or without an hospitalization for SARS-COV-2 infection in the 30 previous days before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 yars
* hip fracture hospitalization
* care code indicating a surgical procedure

Exclusion Criteria:

-Patient with hip fracture hospitalization without a care code indicating a surgical procedure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with hip fracture, and with or without a SARS-COV-2 disease:
  We included all patients older than 65 years with hip fracture hospitalization recorded between March 1, 2020 and December 31, detected through ICD-10 diagnosis codes , and with a DRG Codes (Diagnosis Related Group) indicating a surgical procedure. Patient with hip fracture hospitalization without a care code indicating a surgical procedure were excluded.
  Among these patients, we searched for hospitalizations with SARS-CoV2 diagnostic that occurred within 30 days before the date of hospital admission for hip fracture.
Sampling Method: Non-Probability Sample
Enrollment: 73661 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | Day 0 to Day 30
  hospital mortality within 30 days of the date of hospital admission for hip fracture

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuvillon, Principal Investigator — CHU NIMES
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: No